CLINICAL TRIAL: NCT05879289
Title: Avaliação de eficácia do Efeito Antienvelhecimento de um Suplemento Alimentar na Melhora Das condições da Pele - Estudo Clínico, Subjetivo e Instrumental
Brief Title: Evaluation of the Effectiveness of the Anti-aging Effect of a Supplement in Improving Skin Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Farmoquimica S.A. (Industry)
Collaborators: Medcin Instituto da Pele Ltda (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: EN20-1103
Record Dates: First submitted 2023-05-17; First posted 2023-05-30 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Aging Well
Keywords: dermal aging, elastic fiber, collagen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clinical Trial (Experimental): 36 participants using the product for 90 days. Aims to evaluate the clinical, subjective and instrumental usage
  Interventions: Dietary Supplement: A power supplement

INTERVENTIONS:
Dietary Supplement: A power supplement — A dietary supplement containing vitamins and collagen

SUMMARY:
A unicentric, blind, non-comparative clinical study to evaluate facial and body anti-aging efficacy of a supplement in female participants through clinical, subjective and instrumental evaluations.

DETAILED DESCRIPTION:
A unicentric, blind, non-comparative clinical study to evaluate facial and body anti-aging efficacy of a supplemente in female participants through clinical, subjective and instrumental evaluations.

It will be necessary 33 female participants aged between 35 and 60 years old with signs of aging on the face and neck, complaining of body flaccidity and gynoid lipodystrophy.

The participant will remain in the study for 90 days using the product. Visits will be scheduled in D0, D45 and D90.

Instrumental evaluations: Evaluated on each visit:

* Skin elasticity and firmness using Cutometer - D0, D45 and D90;
* Skin hydration using Corneometer- D0,D45 and D90;
* Detection and accuracy of fine lines and wrinkles using Visia -D0,D45 and D90
* Dermal thickness and density in the thigh region using Ultrasound Voluson E8 before using the product (D0) and after 90 (D90) days of continuous use;
* Participants will respond to a subjective assessment using a questionnaire to capture possible feelings of discomfort during the study and subjective efficacy.
* A dermatologist will be available to monitor the participants throughout the study and respond an assessment of clinical efficiency

ELIGIBILITY:
Inclusion Criteria:

* Signs of aging in the face and neck region (fine lines, furrows and expression lines);
* Participants with complaints of body sagging;
* Participants with BMI < 30 (body mass index less than 30);
* Participants with Gynoid Lipodystrophy Grade 1 and/or 2;
* Agreement to follow the trial procedures and attend the clinic on the days and times determined.
* Ability to understand and consent to their participation in this clinical study, manifested by signing the Term of Free and Informed Consent (TCLE)

Exclusion Criteria:

* Participants who have been diagnosed with COVID-19 by RT-PCR examination or by the presence of IgM antibodies in the serology exam, in the last 4 weeks or who are presenting any of the following symptoms: dry or productive cough, sneezing, runny nose, body ache, headache, anosmia (loss of smell), ageusia (loss of taste) and/or any other symptoms that may be related to covid-19 at the discretion of the investigator;
* Pregnancy or risk of pregnancy/lactation;
* Use of the following topical or systemic medications: immunosuppressants, antihistamines, anti-inflammatories non-hormonal drugs, and corticoids up to 30 days before selection or considering immunosuppressants, the interval should be 3 months before selection;
* Atopic or allergic history to Food Supplements;
* Pathologies and/or active skin lesions (local and/or disseminated) in the assessment area;
* Skin marks in the experimental area that interfere with the evaluation of possible skin reactions (malformations vascular lesions, scars, increased hairiness, large nevus, sunburn);
* Immunosuppression by drugs or active diseases;
* Decompensated endocrinopathies;
* Participants with known congenital or acquired immunodeficiency;
* Relevant medical history or current evidence of alcohol or other drug abuse;
* Known history or suspected intolerance to products of the same category;
* Intense sun exposure up to 15 days before the evaluation;
* Aesthetic or dermatological treatment in the evaluation areas up to 04 weeks before selection;
* Professionals directly involved in carrying out this study;
* Other conditions considered by the evaluating physician as reasonable for disqualification from participation in the study. If so, it should be described under observation in the clinical record

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2022-01-25 (Actual); Primary Completion 2022-05-17 (Actual); Study Completion 2022-05-17 (Actual)

PRIMARY OUTCOMES:
Acceptability in real conditions of use by questionnaire | 90 days
  Evaluate the effectiveness of the investigational product (nutritional supplement) in improving signs of facial and body aging, through clinical, instrumental and subjective evaluations. Confirm in real conditions of use, the absence of risk and irritation and capture feelings of discomfort in the population studied (0 meaning no risk)

SECONDARY OUTCOMES:
Evaluation of skin firmness and elasticity using instrumental evaluation - Cutometer | Day 0, Day 45 e Day 90
  Evaluate the efficacy of the investigational product in improving the firmness and elasticity of the skin through clinical and instrumental evaluations (cutometry) before using the product (D0) and after 45 (D45) and 90 (D90) days of continuous use;
Increase of skin hydration using instrumental evaluation - Corneometer | Day 0, Day 45 e Day 90
  Evaluate the hydration efficacy before using the investigational product D(0) and after 45 (D45) and 90 (D90) days of continuous use through the Corneometer equipment®
Detection and accuracy of fine lines and wrinkles- Visia | Day 0, Day 45 e Day 90
  Evaluate the efficacy of the investigational product in improving wrinkles through instrumental evaluations by Visia® before product use (D0) and after 45 (D45) and 90 (D90) days of use continuous
Increase in dermal thickness and density in the thigh region | Day 0 e Day 90
  Check the increase in dermal thickness and density in the thigh region through Ultrasound Volunson E8 before using the product (D0) and after 90 (D90) days of continuous
Subjective efficacy from the participants | Day 45 e Day 90
  Evaluate the perceived efficacy of the product from the participant's point of view through a subjective questionnaire after 45 (D45) e 90 (D90) days of continuous use of the product
Acceptability in real conditions of use through dermatological questionnaire | Day 0, Day 45 e Day 90
  Check the absence of risk of irritation and capture sensations of discomfort from the studied population, through dermatological evaluation criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Medcin Instituto da Pele, Osasco, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 90 Days